CLINICAL TRIAL: NCT06129864
Title: A Phase III, Randomized, Open-Label, Multi-Center, Global Study of Volrustomig (MEDI5752) as Sequential Therapy Versus Observation in Participants With Unresected Locally Advanced Head and Neck Squamous Cell Carcinoma, Who Have Not Progressed Following Definitive Concurrent Chemoradiotherapy (eVOLVE-HNSCC)
Brief Title: A Global Study of Volrustomig (MEDI5752) for Participants With Unresected Locally Advanced Head and Neck Squamous Cell Carcinoma Following Definitive Concurrent Chemoradiotherapy
Acronym: eVOLVE-HNSCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D798EC00001
Record Dates: First submitted 2023-11-03; First posted 2023-11-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Arm (Experimental): Participants in this arm will receive volrustomig.
  Interventions: Drug: volrustomig
- Observation Arm (No Intervention): Patients in this arm will undergo observation.

INTERVENTIONS:
Drug: volrustomig — volrustomig
  Other Names: MEDI5752
  Arms: Study Arm

SUMMARY:
The main purpose of this study is to assess the efficacy and safety of volrustomig compared to observation in participants with unresected locally advanced head and neck squamous cell carcinoma (LA-HNSCC) who have not progressed after receiving definitive concurrent chemoradiotherapy (cCRT).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced squamous cell carcinoma of the oropharynx, hypopharynx, oral cavity, or larynx with no evidence of metastatic disease (i.e. M0).
* Confirmed unresected Stage III, Stage IVA or IVB according to the eighth edition of the American Joint Committee on Cancer (AJCC) staging manual (tumor, node, metastasis (TNM) staging system).
* Participants will have completed definitive concurrent chemoradiotherapy (cCRT) with curative intent prior to randomization.

Exclusion Criteria:

* Histologically/cytologically confirmed head and neck cancer of any other primary anatomic location in the head and neck not specified in the inclusion criteria including participants with squamous cell carcinoma of unknown primary or non-squamous histologies (eg, nasopharynx or salivary gland). Participants with >1 primary tumors are not eligible for the study.
* Participants with any of the following:

  1. LA-HNSCC that was resected before definitive cCRT
  2. LA-HNSCC that was treated and is recurrent at the time of screening
* Participants who have received radiotherapy (RT) alone as definitive local therapy for LA-HNSCC.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1145 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2028-04-18 (Estimated); Study Completion 2030-09-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) in participants with unresected LA-HNSCC with PD-L1 expressing tumors | Up to approximately 8 years
  PFS is defined as time from randomization until first objective radiological progression per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR), or death due to any cause (in the absence of progression).
  The analysis will include all randomized participants with PD-L1 expressing tumors.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) in the unresected LA-HNSCC intent-to-treat (ITT) population | Up to approximately 8 years
  PFS is defined as time from randomization until first objective radiological progression per RECIST 1.1 as assessed by BICR, or death due to any cause (in the absence of progression).
  The analysis will include all randomized participants.
Landmark Progression-Free Survival (PFS) Rates | Up to approximately 8 years
  PFS is defined as time from randomization until first objective radiological progression per RECIST 1.1 as assessed by BICR, or death due to any cause (in the absence of progression).
  These analyses will include participants with PD-L1 expressing tumors and all randomized participants.
Overall Survival (OS) in participants with unresected LA-HNSCC with PD-L1 expressing tumors | Up to approximately 8 years
  Overall survival (OS) is defined as the time from randomization until the date of death due to any cause.
  The analysis will include all randomized participants with PD-L1 expressing tumors.
Landmark Overall Survival (OS) Rates | Up to approximately 8 years
  OS is defined as the time from randomization until the date of death due to any cause.
  These analyses will include participants with PD-L1 expressing tumors as randomized and all randomized participants.
Overall Survival (OS) in the unresected LA-HNSCC ITT population | Up to approximately 8 years
  OS is defined as the time from randomization until the date of death due to any cause.
  The analysis will include all randomized participants.
Progression Free Survival 2 (PFS2) | Up to approximately 8 years
  PFS2 is defined as the time from randomization until the earliest of the progression event (following the initial investigator-assessed progression), after the start of the first subsequent therapy, or death from any cause, whichever occurs first. The date of the second progression will be recorded by the investigator in the eCRF and defined according to local standard clinical practice.
  These analyses will include participants with PD-L1 expressing tumors as randomized and all randomized participants.
Presence of Anti-Drug-Antibodies (ADAs) against volrustomig in serum | Up to approximately 8 years
  To investigate the immunogenicity of volrustomig.
Participant-reported physical functioning | Up to approximately 8 years
  Change from baseline of physical functioning as measured by scores on the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v.20 - Physical Function 8c are reported on a T score metric (mean = 50 and SD = 10), with higher scores reflecting better physical functioning.
  The analysis will include all randomized participants.
Participant-reported global health status (GHS)/quality of life (QoL) | Up to approximately 8 years
  Change from baseline of Global Health Status/Quality of Life subscale scores as measured by the European Organization for Research and Treatment of Cancer (EORTC) Item Library 172 are transformed to a 0-100 range; a higher score represents higher quality of life.
  The analysis will include all randomized participants.
Percentage of participants with Adverse Events | Up to approximately 8 years
  Adverse Events as assessed by Common Terminology Criteria for Adverse Events (CTCAE).
Area under the curve (AUC) | Up to approximately 8 years
  The concentration of Volrustomig in serum will be determined. Area under the curve is the integral of the concentration-time curve. The AUC reflects the actual body exposure to drug after administration. The AUC is dependent on the rate of elimination of the drug from the body and the dose administered.
Maximum plasma concentration of the drug (Cmax) | Up to approximately 8 years
  The concentration of Volrustomig in serum will be determined (Cmax will be derived).
The time taken to reach the maximum concentration (Tmax) | Up to approximately 8 years
  The concentration of Volrustomig in serum will be determined (Tmax will be derived).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Haddad, MD, Study Chair — Dana Farber Cancer Institute Massachusetts, USA; Lisa Licitra, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori and University of Milan Milan, Italy
Locations (263):
- United States (64):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Prescott Valley, Arizona
  - Research Site, Springdale, Arkansas
  - Research Site, Fountain Valley, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Santa Rosa, California
  - Research Site, Whittier, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Lone Tree, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Myers, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Palm Bay, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Niles, Illinois
  - Research Site, Des Moines, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Hyattsville, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Upper Marlboro, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Fairhaven, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, East Brunswick, New Jersey
  - Research Site, Hackensack, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Flower Mound, Texas
  - Research Site, Houston, Texas
  - Research Site, Odessa, Texas
  - Research Site, Tyler, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, West Jordan, Utah
  - Research Site, Fairfax, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
- Austria (5):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (5):
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Jette
  - Research Site, La Louvière
  - Research Site, Namur
- Brazil (12):
  - Research Site, Barretos
  - Research Site, Florianópolis
  - Research Site, Fortaleza
  - Research Site, Ijuí
  - Research Site, Ipatinga
  - Research Site, Londrina
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
  - Research Site, Teresina
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Regina
- China (30):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dongwan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Huizhou
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Zhengzhou
  - Research Site, Zhuhai
- France (8):
  - Research Site, Avignon
  - Research Site, Bordeaux
  - Research Site, Le Mans
  - Research Site, Lyon
  - Research Site, Nice
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (14):
  - Research Site, Berlin
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Greifswald
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, München
  - Research Site, Rostock
  - Research Site, Tübingen
  - Research Site, Ulm
  - Research Site, Würzburg
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szekszárd
- India (14):
  - Research Site, Bengaluru
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kanpur
  - Research Site, Kochi
  - Research Site, Kolkata
  - Research Site, Lucknow
  - Research Site, Madurai
  - Research Site, Mohali
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Thiruvananthapuram
  - Research Site, Vadodara
  - Research Site, Varanasi
- Italy (8):
  - Research Site, Aviano
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Rozzano
- Japan (21):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hidaka-shi
  - Research Site, Hiroshima
  - Research Site, Kashiwa
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Shiwa-gun
  - Research Site, Sunto-gun
  - Research Site, Yokohama
- Malaysia (5):
  - Research Site, George Town
  - Research Site, Johor Bahru
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Kuching
- Philippines (7):
  - Research Site, Cebu City
  - Research Site, General Santos
  - Research Site, Iloilo City
  - Research Site, Manila
  - Research Site, Pasig
  - Research Site, Quezon City
  - Research Site, West San Juan City
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Gliwice
  - Research Site, Olsztyn
  - Research Site, Piotrkow Trybunalski
  - Research Site, Siedlce
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
- Research Site, San Juan, Puerto Rico
- South Korea (5):
  - Research Site, Goyang-si
  - Research Site, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (5):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Jaén
  - Research Site, Madrid
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (7):
  - Research Site, Bangkok
  - Research Site, Chaing Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Lampang
  - Research Site, Muang
  - Research Site, Mueang
- Turkey (Türkiye) (6):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Eskişehir
  - Research Site, Istanbul
  - Research Site, Karşıyaka
  - Research Site, Yenimahalle
- United Kingdom (10):
  - Research Site, Aberdeen
  - Research Site, Cambridge
  - Research Site, Hampshire
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Northwood
  - Research Site, Sutton
  - Research Site, Taunton
- Vietnam (6):
  - Research Site, Da Nang
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Huế
  - Research Site, Vinh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles.
  For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool .
  Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
  Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home